CLINICAL TRIAL: NCT06646809
Title: Reducing Inflammatory Syndrome in Surgery - Colorectal (RISIS-CR) Trial
Acronym: RISIS-CR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/00724
Record Dates: First submitted 2023-07-24; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Geroprotector; Alpha-ketoglutarate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ketoglutaric Acids; Standard of Care

STUDY DESIGN:
Intervention Model Description: 3 groups of patients - low inflammatory responder, high inflammatory responder with AKG, high inflammatory responder with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low inflammatory responder (Other): Low inflammatory responder group - to receive standard care
  Interventions: Other: Standard care
- High inflammatory responder - AKG (Experimental): High inflammatory responder group - to receive AKG tablets (1g a day, once a day, taken orally)
  Interventions: Dietary Supplement: Alpha-ketoglutarate
- High inflammatory responder - placebo (Placebo Comparator): High inflammatory responder group - to receive placebo tablets (1g a day, once a day, taken orally)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-ketoglutarate — Alpha-ketoglutarate supplements
  Arms: High inflammatory responder - AKG
Dietary Supplement: Placebo — Placebo tablets
  Arms: High inflammatory responder - placebo
Other: Standard care — Standard care
  Arms: Low inflammatory responder

SUMMARY:
The study proposes to identify inflammatory responsiveness of patients prior to CRC surgery and administer prophylactic anti-inflammatory treatment targeted only to those with an excessive pro-inflammatory response. The study team believe this to be a creative approach as the principles of personalized medicine will be used to treat the appropriate patients, and equally as importantly, to not further suppress the inflammatory response of those who have poor immune function already.

Geroprotectors reduce inflammation, and may reduce postoperative SIR and complications after CRC surgery. In this proposal, we intend to use alpha ketoglutarate (AKG), a geroprotector supplement that enjoys a GRAS (generally regarded as safe) status with the FDA. [12] Apart from reducing inflammation and inhibiting the mTOR pathway, AKG also prevents loss of muscle mass, improves brain oxygenation, has cardioprotective effects, and improves renal function. It also has anti-cancer effects beyond mTOR pathway inhibition, including regulating HIF-1 activity, suppressing secretion of angiogenic factors, and regulating epigenetic processes.

DETAILED DESCRIPTION:
The incidence of colorectal cancer (CRC) increases exponentially with age, with >50% of CRC first diagnosed at 50 years or older. Surgery is the mainstay of treatment. However, older patients are more likely to develop postoperative ileus and anastomotic leak, longer hospital stays and higher mortality. In the long-term, they are more likely to experience fatigue and slow recovery.

Surgery triggers an inflammatory response. In some cases, the immune system is unable to distinguish between the stimuli of major surgery (ideally a modest response) and trauma or infection. This overshoot manifests as a postoperative systemic inflammatory response (SIR) and may lead to tissue destruction and organ dysfunction. In CRC surgery, SIR as defined by C-reactive protein (CRP) elevation is associated with postoperative Clavien-Dindo grades III and IV complications where intervention is needed. These complications include infection and anastomotic leak, and are linked to reduced overall survival independent of both surgery-related complications and tumour stage. In addition, preoperative systemic inflammation is a marker of poor prognosis. As ageing is often accompanied by a chronic low-grade inflammation, it was not surprising that preoperative systemic inflammation is more common in older patients.

The use of anti-inflammatory drugs to reduce SIR has had mixed successes. Chronic steroid use is a recognized risk factor for anastomotic leak, but in a recent meta-analysis, the use of preoperative corticosteroids lowered markers of SIR and reduced postoperative infective complications. Similarly, although NSAIDs have been shown to reduce hospital stay and hasten recovery in bowel function, a recent meta-analysis indicated that it increases the risk of anastomotic leaks.

Older patients may have impaired immune response to surgical stress from immunosenescence but conversely, some may develop a more intense and prolonged response. In a population study of elderly people, this heterogeneity conferred a survival benefit to those who could mount a pro-inflammatory response, whereas those with poor pro-inflammatory response were more prone to infections. Therefore, suppressing the postoperative SIR in pro-inflammatory patients is likely beneficial but not in patients with low pro-inflammatory potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 45 years old
* Undergoing elective colorectal cancer surgery
* Able to give informed consent

Exclusion Criteria:

* Undergoing emergency colorectal cancer surgery
* Unable to give informed consent
* Females who are pregnant
* Cognitively impaired patients

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of postoperative CRP levels between the low inflammatory responders, high inflammatory responders with AKG and high inflammatory responders with placebo | Postoperative till day 30
  Comparison of postoperative CRP levels between the groups.

SECONDARY OUTCOMES:
Compare changes in frailty, cognition, recovery trajectory, clinical outcomes, and surgical complications | Postoperative till day 30
  Compare changes in frailty, cognition, recovery trajectory, clinical outcomes, and surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Hospital, Singapore
Locations (4):
- Singapore (4):
  - National University Hospital, Singapore, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No